CLINICAL TRIAL: NCT00745056
Title: Women's Health Initiative Memory Study--Epidemiology of Cognitive Health Outcomes
Brief Title: Examining the Relationship Between Hormone Therapy (HT) and Cognitive Function (The WHIMS-ECHO Study)
Acronym: WHIMS-ECHO
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: BG04-310
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2021-04

CONDITIONS: Dementia
Keywords: Cognition; Memory; Hormone Therapy; HT
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective, observational study of the cohort of older post-menopausal participants in the WHI Memory Study, a sub-cohort of participants in the WHI Hormone Trials. Annual cognitive assessments and ascertainment of cognitive impairment enable the continued monitoring of long-term effects of randomization to HT on cognition and identification of predictors of cognitive vulnerability and resilience in older women.

DETAILED DESCRIPTION:
Identification of the predictors of cognitive impairment and cognitive resilience among aging women is important because the incidence of mild cognitive impairment (MCI) and dementia increases with age and women live the longest. The Women's Health Initiative Memory Study examined the impact of randomization to hormone therapy (conjugated equine estrogen alone or in combination with medroxyprogesterone vs. placebo) in a subset of participants aged 65-79 years at enrollment into WHI and the WHI Hormone Trials. WHIMS revealed an increased risk of all-cause dementia and MCI plus poorer global cognitive function among women randomized to HT compared to those receiving placebo. WHIMS ECHO is a prospective, observational study of the remaining cohort of WHIMS participants following cessation of treatment. Annual cognitive assessments of learning, attention, memory, working memory, executive function and language are conducted by telephone by trained staff and adjudication of incident cognitive impairment (MCI and dementia) continues. This enables the continued monitoring of long-term effects of randomization to HT on cognition and identification of predictors of cognitive aging and resilience in older women.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the WHIMS study

Exclusion Criteria

* Non-English speaking
* Hearing Impaired

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants will include women who participated in the WHIMS study.
Sampling Method: Probability Sample
Enrollment: 2922 (Actual)
Dates: Start 2008-09-11 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
All-cause dementia and Mild Cognitive Impairment | Measured annually

SECONDARY OUTCOMES:
Global and domain specific cognitive function | Measured annually

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Rapp, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
WHIMS-ECHO will follow guidelines, methods and processes as set forth in the WHI 2015-2020 Data Sharing Plan. Limited data sets will be archived on the WHIMS-ECHO website. Accompanying the limited data sets, substantial electronic documentation will be provided in a standard format that is readable on a variety of platforms. Documentation will include data collection forms, a description of study protocol and procedures, description of all variable re-coding and a list of major study publications. These data will be available to users only under a data-sharing agreement that provides for: a commitment to using the data only for research purposes and not to identify any individual participant; a commitment to securing the data using appropriate computer technology; and a commitment to destroying or returning the data after analyses are completed. Data will be made available for timely release no later than the acceptance for publication of the main findings from the final dataset.

REFERENCES:
- [Background] Shumaker SA, Legault C, Rapp SR, Thal L, Wallace RB, Ockene JK, Hendrix SL, Jones BN 3rd, Assaf AR, Jackson RD, Kotchen JM, Wassertheil-Smoller S, Wactawski-Wende J; WHIMS Investigators. Estrogen plus progestin and the incidence of dementia and mild cognitive impairment in postmenopausal women: the Women's Health Initiative Memory Study: a randomized controlled trial. JAMA. 2003 May 28;289(20):2651-62. doi: 10.1001/jama.289.20.2651. PMID 12771112
- [Background] Vaughan L, Erickson KI, Espeland MA, Smith JC, Tindle HA, Rapp SR. Concurrent and longitudinal relationships between cognitive activity, cognitive performance, and brain volume in older adult women. J Gerontol B Psychol Sci Soc Sci. 2014 Nov;69(6):826-36. doi: 10.1093/geronb/gbu109. Epub 2014 Sep 10. PMID 25209372
- [Background] Gaussoin SA, Espeland MA, Absher J, Howard BV, Jones BM, Rapp SR. Ascertaining dementia-related outcomes for deceased or proxy-dependent participants: an overview of the Women's Health Initiative Memory Study supplemental case ascertainment protocol. Int J Geriatr Psychiatry. 2012 Feb;27(2):205-14. doi: 10.1002/gps.2714. Epub 2011 Mar 18. PMID 21416508
- [Background] Voytko ML. Women's cognitive health special edition. Age (Dordr). 2009 Sep;31(3):189-90. doi: 10.1007/s11357-009-9090-7. Epub 2009 Mar 10. No abstract available. PMID 19277900
- [Result] Vaughan L, Leng I, Dagenbach D, Resnick SM, Rapp SR, Jennings JM, Brunner RL, Simpson SL, Beavers DP, Coker LH, Gaussoin SA, Sink KM, Espeland MA. Intraindividual variability in domain-specific cognition and risk of mild cognitive impairment and dementia. Curr Gerontol Geriatr Res. 2013;2013:495793. doi: 10.1155/2013/495793. Epub 2013 Dec 22. PMID 24454359
- [Result] Haring B, Leng X, Robinson J, Johnson KC, Jackson RD, Beyth R, Wactawski-Wende J, von Ballmoos MW, Goveas JS, Kuller LH, Wassertheil-Smoller S. Cardiovascular disease and cognitive decline in postmenopausal women: results from the Women's Health Initiative Memory Study. J Am Heart Assoc. 2013 Dec 18;2(6):e000369. doi: 10.1161/JAHA.113.000369. PMID 24351701
- [Result] Rossom RC, Espeland MA, Manson JE, Dysken MW, Johnson KC, Lane DS, LeBlanc ES, Lederle FA, Masaki KH, Margolis KL. Calcium and vitamin D supplementation and cognitive impairment in the women's health initiative. J Am Geriatr Soc. 2012 Dec;60(12):2197-205. doi: 10.1111/jgs.12032. Epub 2012 Nov 23. PMID 23176129
- [Result] Goveas JS, Hogan PE, Kotchen JM, Smoller JW, Denburg NL, Manson JE, Tummala A, Mysiw WJ, Ockene JK, Woods NF, Espeland MA, Wassertheil-Smoller S. Depressive symptoms, antidepressant use, and future cognitive health in postmenopausal women: the Women's Health Initiative Memory Study. Int Psychogeriatr. 2012 Aug;24(8):1252-64. doi: 10.1017/S1041610211002778. Epub 2012 Feb 3. PMID 22301077
- [Result] Haan M, Espeland MA, Klein BE, Casanova R, Gaussoin SA, Jackson RD, Millen AE, Resnick SM, Rossouw JE, Shumaker SA, Wallace R, Yaffe K; Women's Health Initiative Memory Study and the Women's Health Initiative Sight Exam. Cognitive function and retinal and ischemic brain changes: the Women's Health Initiative. Neurology. 2012 Mar 27;78(13):942-9. doi: 10.1212/WNL.0b013e31824d9655. Epub 2012 Mar 14. PMID 22422889
- [Result] Shih RA, Ghosh-Dastidar B, Margolis KL, Slaughter ME, Jewell A, Bird CE, Eibner C, Denburg NL, Ockene J, Messina CR, Espeland MA. Neighborhood socioeconomic status and cognitive function in women. Am J Public Health. 2011 Sep;101(9):1721-8. doi: 10.2105/AJPH.2011.300169. Epub 2011 Jul 21. PMID 21778482
- [Result] Goveas JS, Espeland MA, Woods NF, Wassertheil-Smoller S, Kotchen JM. Depressive symptoms and incidence of mild cognitive impairment and probable dementia in elderly women: the Women's Health Initiative Memory Study. J Am Geriatr Soc. 2011 Jan;59(1):57-66. doi: 10.1111/j.1532-5415.2010.03233.x. PMID 21226676
- [Result] Kerwin DR, Gaussoin SA, Chlebowski RT, Kuller LH, Vitolins M, Coker LH, Kotchen JM, Nicklas BJ, Wassertheil-Smoller S, Hoffmann RG, Espeland MA; Women's Health Initiative Memory Study. Interaction between body mass index and central adiposity and risk of incident cognitive impairment and dementia: results from the Women's Health Initiative Memory Study. J Am Geriatr Soc. 2011 Jan;59(1):107-12. doi: 10.1111/j.1532-5415.2010.03219.x. PMID 21226681
- [Result] Rapp SR, Legault C, Henderson VW, Brunner RL, Masaki K, Jones B, Absher J, Thal L. Subtypes of mild cognitive impairment in older postmenopausal women: the Women's Health Initiative Memory Study. Alzheimer Dis Assoc Disord. 2010 Jul-Sep;24(3):248-55. doi: 10.1097/WAD.0b013e3181d715d5. PMID 20473134
- [Result] Atkinson HH, Rapp SR, Williamson JD, Lovato J, Absher JR, Gass M, Henderson VW, Johnson KC, Kostis JB, Sink KM, Mouton CP, Ockene JK, Stefanick ML, Lane DS, Espeland MA. The relationship between cognitive function and physical performance in older women: results from the women's health initiative memory study. J Gerontol A Biol Sci Med Sci. 2010 Mar;65(3):300-6. doi: 10.1093/gerona/glp149. Epub 2009 Sep 29. PMID 19789197
- [Result] Coker LH, Espeland MA, Rapp SR, Legault C, Resnick SM, Hogan P, Gaussoin S, Dailey M, Shumaker SA. Postmenopausal hormone therapy and cognitive outcomes: the Women's Health Initiative Memory Study (WHIMS). J Steroid Biochem Mol Biol. 2010 Feb 28;118(4-5):304-10. doi: 10.1016/j.jsbmb.2009.11.007. Epub 2009 Nov 22. PMID 19932751
- [Result] Colenda CC, Legault C, Rapp SR, DeBon MW, Hogan P, Wallace R, Hershey L, Ockene J, Whitmer R, Phillips LS, Sarto GE. Psychiatric disorders and cognitive dysfunction among older, postmenopausal women: results from the Women's Health Initiative Memory Study. Am J Geriatr Psychiatry. 2010 Feb;18(2):177-86. doi: 10.1097/JGP.0b013e3181c65864. PMID 20104074
- [Result] Espeland MA, Tindle HA, Bushnell CA, Jaramillo SA, Kuller LH, Margolis KL, Mysiw WJ, Maldjian JA, Melhem ER, Resnick SM; Women's Health Initiative Memory Study. Brain volumes, cognitive impairment, and conjugated equine estrogens. J Gerontol A Biol Sci Med Sci. 2009 Dec;64(12):1243-50. doi: 10.1093/gerona/glp128. Epub 2009 Sep 3. PMID 19729392
- [Result] Chen JC, Brunner RL, Ren H, Wassertheil-Smoller S, Larson JC, Levine DW, Allison M, Naughton MJ, Stefanick ML. Sleep duration and risk of ischemic stroke in postmenopausal women. Stroke. 2008 Dec;39(12):3185-92. doi: 10.1161/STROKEAHA.108.521773. Epub 2008 Jul 17. PMID 18635832
- [Result] Johnson KC, Margolis KL, Espeland MA, Colenda CC, Fillit H, Manson JE, Masaki KH, Mouton CP, Prineas R, Robinson JG, Wassertheil-Smoller S; Women's Health Initiative Memory Study and Women's Health Initiative Investigators. A prospective study of the effect of hypertension and baseline blood pressure on cognitive decline and dementia in postmenopausal women: the Women's Health Initiative Memory Study. J Am Geriatr Soc. 2008 Aug;56(8):1449-58. doi: 10.1111/j.1532-5415.2008.01806.x. Epub 2008 Jul 15. PMID 18637980
- [Derived] Haring B, Wu C, Coker LH, Seth A, Snetselaar L, Manson JE, Rossouw JE, Wassertheil-Smoller S. Hypertension, Dietary Sodium, and Cognitive Decline: Results From the Women's Health Initiative Memory Study. Am J Hypertens. 2016 Feb;29(2):202-16. doi: 10.1093/ajh/hpv081. Epub 2015 Jul 1. PMID 26137952